CLINICAL TRIAL: NCT00467571
Title: Helicobacter Pylori Infection in Children With Chronic Idiopathic Thrombocytopenic Purpura
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Ramathibodi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID11-48-20
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2008-09

CONDITIONS: Chronic Idiopathic Thrombocytopenic Purpura; Helicobacter Pylori Infection
Keywords: chronic idiopathic thrombocytopenic purpura; Helicobacter pylori infection; platelet
MeSH Terms: interventions — Lansoprazole; Clarithromycin; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental): Drug: lansoprazole, clarithromycin, amoxycillin
  Interventions: Drug: lansoprazole, clarithromycin, amoxycillin

INTERVENTIONS:
Drug: lansoprazole, clarithromycin, amoxycillin — lansoprazole (15, 30 mg) 1 tab twice daily, clarithromycin 7.5 mg/kg twice daily, amoxycillin 25 mg/kg twice daily; rout: orally; duration 14 days
  Other Names: lansoprazole or Prevacid; clarithromycin or Klacid; Amoxycillin or Ibiamox

SUMMARY:
Previous studies suggest that chronic idiopathic thrombocytopenic purpura is associated with Helicobacter pylori infection. The objective is to study the effect of Helicobacter pylori eradication on platelet count.

DETAILED DESCRIPTION:
Children with chronic idiopathic thrombocytopenic purpura who have Helicobacter pylori infection are enrolled. Helicobacter pylori infection is diagnosed by urea breath test. Patients who have Helicobacter pylori infection will be randomized into 2 groups: control and treatment groups. The treatment group will receive 2 antibiotics and proton-pump inhibitors for 14 days for eradication of infection. Repeated urea breath test at week 6-8 after treatment. Blood tests for platelet count will be performed every month for 6 months in both groups. Platelet count at 6 months in both group will be compared.Blood for platelet antibody will be performed at 3 and 6 months. Control group will receive treatment for Helicobacter pylori at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Children who was diagnosed as chronic ITP, defined by platelets below 100,000/uL for more than 6 months without identified causes.
* 13C-urea breath test (UBT) was performed for diagnosis of Helicobacter pylori infection.

Exclusion Criteria:

* Patients who had a previous treatment for H. pylori infection.

  * Patients require prednisolone more than 0.5 mg/kg/day

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2006-03; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
platelet count | 6 months

SECONDARY OUTCOMES:
platelet antibody after treatment of Helicobacter pylori infection, compared with control group (no treatment of Helicobacter pylori) | 6 months
platelet count | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Suporn Treepongkaruna, M.D., Principal Investigator — Ramathibodi Hospital
Locations (1):
- Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Bangkok, Bangkok, Thailand